CLINICAL TRIAL: NCT03413904
Title: Transanal Versus Laparoscopic Total Mesorectal Excision For Mid And Low Rectal Cancer. A Multicentre Randomised Clinical Trial on Anastomotic Leak
Brief Title: Transanal Versus Laparoscopic Total Mesorectal Excision for Rectal Cancer.
Acronym: taTME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, vignali andrea, Professor, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: taTME
Record Dates: First submitted 2018-01-15; First posted 2018-01-29 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Rectal Cancer
Keywords: taTME
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transanal TME (Experimental): Study procedure will consist in 2-team (combined) LAR with transanal TME using laparoscopic abdominal assistance.Transanal TME is performed either at the same time or following the above steps. Transanal endoscopic TME dissection will proceed circumferentially until the peritoneal cavity is entered anteriorly. Following complete mobilization of the rectosigmoid, the specimen is extracted transanally or using a Pfannenstiel incision followed by colorectal anastomosis, and a temporary diverting stoma will be created, which is standard of care following surgery for this type of cancer.
  Interventions: Procedure: transanal TME
- laparoscopic TME (Active Comparator): Procedure will consist in 1 team performing laparoscopic TME. Following stapled closure of the rectum below the tumor, and complete mobilization of the rectosigmoid, the specimen is extracted using a Pfannenstiel incision . A stapled (knight-Griffen) colorectal anastomosis or coloanal anastomosis will be created and a temporary diverting stoma will be fashioned which is standard of care following surgery for this type of cancer.
  Interventions: Procedure: laparoscopic TME

INTERVENTIONS:
Procedure: transanal TME — transanal approach to TME in rectal cancer
  Arms: transanal TME
Procedure: laparoscopic TME — laparoscopic approach to TME in rectal cancer
  Arms: laparoscopic TME

SUMMARY:
This study is designed as a prospective, multi-center, randomized, open-labelled, parallel group, non-inferiority trial. The aim of this study is to evaluate the TaTME technique compared with conventional laparoscopic rectal surgery, focusing on, anastomotic dehiscence, conversion rate to open surgery, hospital stay and long-term functional outcomes.

DETAILED DESCRIPTION:
This study is designed as a prospective, multi-center, randomized, open-labelled, parallel group, non-inferiority trial. The patients will be randomized and assigned to transanal mesorectal excision (TaTME) or laparoscopic mesorectal excision (LpTME) at a ratio 1:1, based on a centralized computer generated, blocked randomization list stratified by center. Six centers will be involved. Within each center a block size of four will be used, stratified by gender and age (±3 years). A central electronic data capture system will be generated by the promoting center for data collection. All the participating surgeons and centers will be required to document their previous experience with TaTME (a minimum of 10 documented procedures is required). Moreover, they will be invited to submit a video showing their surgical technique in performing a TaTME operation (said video must contain no reference to patient ID, and is used exclusively to demonstrate the participating surgeon's technique). The video will be reviewed by the promoting center in order to standardize the procedure, prior to the beginning of the recruitment process. In each center, before starting effective recruitment of patients to the trial, the surgical team will be required to perform a minimum of 4 TaTME operations based on the adopted standardized procedure to calibrate the participant surgeons.

All statistical analyses will be conducted on an "intention to treat" basis.

Statistical methodology The trial is designed as a non-inferiority trial. In statistical terms, the study will establish whether the anastomotic rate (%) for the experimental treatment is not worse than the anastomotic rate (%) for the standard treatment by more than a specific non-inferiority margin, δ, set to 0.05, with δ denoting the difference anastomotic rate rates (experimental vs. control). Formally, the study will test the one-sided null hypothesis H0: δ > = 5% vs. the alternative H1: δ < 5%, and will reject the null hypothesis with a 5% level of significance if the upper bound of a standard asymptotic 90% confidence interval for difference in proportions is below the 5% non-inferiority margin.

Sample size In recent studies (1-5) estimating the anastomotic leak ("failure") rate (%) in the standard LpTME (control technique) ranged from 6.4 to 18.8 % (median of studies, 13%), while in the two recent studies evaluating TaTME (experimental technique) it was 6.7% and 8.6 %, respectively, (resulting in a weighted rate of 7%). The investigators therefore hypothesised a failure rate of 13% (that equivalently means a "success" rate of 87%) in the control arm and a crude (relative) 6% (4.6%) reduction in the experimental arm (that equivalently means a "success" rate of 93%) over the standard arm. Based on the non-inferiority hypothesis and the above findings, and assuming a non-inferiority limit of 0.05, a total of 184 patients (92 for each arm) is required i.e., if there is a true difference in favour of the experimental treatment of 6%, then 184 patients are required to be 80% sure that the upper limit of a one-sided 95% confidence interval (or equivalently a 90% two-sided confidence interval) will exclude a difference in favour of the standard group of more than 5%. The inclusion period will be of 2 years. The results will be available within 3 years of starting recruitment. The investigators will consider still acceptable and not different clinically a failure rate of 18% (i.e., a non-inferiority limit of 5%) as this value is below the 18.8% maximum failure rate estimated in the standard LpTME. Additionally, the non-inferiority limit of 5% has been also recently indicated in a similar trial (ETAP-GRECCAR 11 TRIAL) (assuming conversion to open as "failure" event) registered at clinicalTrials.gov, NCT02584985.

Statistical analysis Both per-protocol and intention-to-treat analysis will be performed, as currently recommended in literature. Descriptive data for continuous variables will be reported as mean (standard deviation [SD]) or median (25th and 75th percentiles), as appropriate. Descriptive data for categorical variables will be reported as number of observations (percentage). For continuous variables, univariate comparison between LpTME and TaTME will be performed by the Student's t test for normally distributed data (based on the Kolmogorov-Smirnov test) or the Mann-Whitney U test for non-normally distributed data. The chi-square test, or the Fisher exact test, as well the Kruskal-Wallis test, as appropriate, will be used for comparing discrete variables. Logistic regression models will be additionally carried out and survival analysis of postoperative binary outcomes, as appropriate. All the statistical tests will be performed by using the SPSS statistical package, version 20.0 (SPSS Inc., Chicago, IL) for Windows (Microsoft, Redmond, WA).

Study procedure:

Study procedures will consist in 2-team (combined) low anterior resection with transanal TME using laparoscopic abdominal assistance. Laparoscopic abdominal access will be obtained followed by inferior mesenteric vessels transection, mobilization of the proximal colon and splenic flexure takedown will be performed in all cases. Transanal TME is performed either at the same time or following the above steps. Following pursestring closure of the rectum below the tumor, transanal endoscopic TME dissection will proceed circumferentially until the peritoneal cavity is entered anteriorly. Following complete mobilization of the rectosigmoid, the specimen will be extracted transanally or using a Pfannenstiel incision followed by colorectal anastomosis, and a temporary diverting stoma will be created, which is standard of care following surgery for this type of cancer. At the end of the surgical procedure a macroscopical examination of the specimen will be conducted by the surgeon in conjunction with the pathologist.

Postoperative care and follow-up:

All patients enrolled in the study will be managed according to same standard postoperative protocols. Postoperative visits and oncology follow-up visits will occur as per standard practice and oncologic outcomes. The duration of postoperative follow up for each patient will be 3 years.

DATA OWNERSHIP AND PUBLICATION

The single participating centers will gather the data which will then be analyzed centrally by the promoting center. The promoting center will aim to publish said data in an adequate scientific journal and share the results with the principal investigators (PIs) of all participating centers.

ADVERSE EVENTS

All adverse events will be notified to the promoting centre by Case Report File (CRF). The promoting center will then gather the data and promptly notify the PIs and Ethic Committees of all participating centers.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven solitary mid and low rectal cancer
* proven by rigid rectoscopy, pelvic MRI and digital rectal examination (DRE)
* amenable to curative sphincter-preserving surgery
* no evidence of distant metastases (T3-4a,N0 or T1-4a,N1-2)
* if evaluated after neoadiuvant therapy, no evidence of threaten of the mesorectal fascia (MRF) after therapy

Exclusion Criteria:

* no indication to perform sphincter preservation surgery (Tumors invading into the internal anal sphincter muscle based on pelvic MRI)
* T4b tumor invading adjacent organs
* recurrent cancer
* concurrent or previous diagnosis of invasive cancer within 5 years
* prior history of colorectal resection
* tumors with in growth more than 1/3 of anal sphincter complex or levator ani.
* presence of fecal incontinence at baseline according to Wexner's classification
* emergent surgery with intestinal obstruction or perforation
* absolute contraindications to general anaesthesia or prolonged pneumoperitoneum, such as severe cardiovascular or respiratory disease (ASA class > III)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2018-03-27 (Actual); Primary Completion 2020-02-29 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Anastomotic leakage | 30 days
  Evaluate the effectiveness of the T-TME versus L-LAR in term of clinically evident anastomotic leak rate.
Conversion to open | intraoperative
  Evaluate the effectiveness of the T-TME versus L-LAR in term of conversion to open surgery

SECONDARY OUTCOMES:
Pathology | 30 days
  Complete pathology assessment of TME specimens according to Quirke classification
QoL | 12 months
  Evaluate the effectiveness of the T-TME versus L-LAR on quality of life assessed with Short-Form Health Survey (SF-36) score in patients with rectal cancer. The questionnaire consists of eight sections, each of which is evaluated 0 (most disability) to 100 (least disability).
Functional results | 12 months
  Evaluating functional results after ileostomy closure. The evaluation will be done using the Fecal Incontinence Quality of Life Questionnaire (FIQL). Scales range from 1 to 4; with a 1 indicating a lower functional status of quality of life. Scales scores are the average (mean) response to all items in the scale.
Functional results 2 | 12 months
  Evaluating functional results after ileostomy closure.The evaluation will be done using Wexner scores (range 0-20 i.e. least-most incontinence) in patients with rectal cancer.
postoperative complications | 30 days
  evaluating postoperative complications after surgery according to Clavien-Dindo Classification
Long-term postoperative complications | 36 months
  evaluating long-term postoperative complications following hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Vignali, Principal Investigator — IRCCS San Raffaele
Locations (1):
- IRCCS San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kang J, Choi GS, Oh JH, Kim NK, Park JS, Kim MJ, Lee KY, Baik SH. Multicenter Analysis of Long-Term Oncologic Impact of Anastomotic Leakage After Laparoscopic Total Mesorectal Excision: The Korean Laparoscopic Colorectal Surgery Study Group. Medicine (Baltimore). 2015 Jul;94(29):e1202. doi: 10.1097/MD.0000000000001202. PMID 26200636
- [Background] Leroy J, Jamali F, Forbes L, Smith M, Rubino F, Mutter D, Marescaux J. Laparoscopic total mesorectal excision (TME) for rectal cancer surgery: long-term outcomes. Surg Endosc. 2004 Feb;18(2):281-9. doi: 10.1007/s00464-002-8877-8. Epub 2003 Dec 29. PMID 14691716
- [Background] Morino M, Parini U, Giraudo G, Salval M, Brachet Contul R, Garrone C. Laparoscopic total mesorectal excision: a consecutive series of 100 patients. Ann Surg. 2003 Mar;237(3):335-42. doi: 10.1097/01.SLA.0000055270.48242.D2. PMID 12616116
- [Background] Goldberg S, Klas JV. Total mesorectal excision in the treatment of rectal cancer: a view from the USA. Semin Surg Oncol. 1998 Sep;15(2):87-90. doi: 10.1002/(sici)1098-2388(199809)15:23.0.co;2-1. PMID 9730414
- [Background] Kapiteijn E, Kranenbarg EK, Steup WH, Taat CW, Rutten HJ, Wiggers T, van Krieken JH, Hermans J, Leer JW, van de Velde CJ. Total mesorectal excision (TME) with or without preoperative radiotherapy in the treatment of primary rectal cancer. Prospective randomised trial with standard operative and histopathological techniques. Dutch ColoRectal Cancer Group. Eur J Surg. 1999 May;165(5):410-20. doi: 10.1080/110241599750006613. PMID 10391155
- [Background] Marks JH, Myers EA, Zeger EL, Denittis AS, Gummadi M, Marks GJ. Long-term outcomes by a transanal approach to total mesorectal excision for rectal cancer. Surg Endosc. 2017 Dec;31(12):5248-5257. doi: 10.1007/s00464-017-5597-7. Epub 2017 Jun 22. PMID 28643051
- [Background] Arroyave MC, DeLacy FB, Lacy AM. Transanal total mesorectal excision (TaTME) for rectal cancer: Step by step description of the surgical technique for a two-teams approach. Eur J Surg Oncol. 2017 Feb;43(2):502-505. doi: 10.1016/j.ejso.2016.10.024. Epub 2016 Nov 20. PMID 27914773
- [Background] Penna M, Hompes R, Arnold S, Wynn G, Austin R, Warusavitarne J, Moran B, Hanna GB, Mortensen NJ, Tekkis PP; TaTME Registry Collaborative. Transanal Total Mesorectal Excision: International Registry Results of the First 720 Cases. Ann Surg. 2017 Jul;266(1):111-117. doi: 10.1097/SLA.0000000000001948. PMID 27735827
- [Background] Atallah S, Albert M, Monson JR. Critical concepts and important anatomic landmarks encountered during transanal total mesorectal excision (taTME): toward the mastery of a new operation for rectal cancer surgery. Tech Coloproctol. 2016 Jul;20(7):483-94. doi: 10.1007/s10151-016-1475-x. Epub 2016 May 17. PMID 27189442
- [Background] Deijen CL, Velthuis S, Tsai A, Mavroveli S, de Lange-de Klerk ES, Sietses C, Tuynman JB, Lacy AM, Hanna GB, Bonjer HJ. COLOR III: a multicentre randomised clinical trial comparing transanal TME versus laparoscopic TME for mid and low rectal cancer. Surg Endosc. 2016 Aug;30(8):3210-5. doi: 10.1007/s00464-015-4615-x. Epub 2015 Nov 4. PMID 26537907
- [Background] Lacy AM, Adelsdorfer C, Delgado S, Sylla P, Rattner DW. Minilaparoscopy-assisted transrectal low anterior resection (LAR): a preliminary study. Surg Endosc. 2013 Jan;27(1):339-46. doi: 10.1007/s00464-012-2443-9. Epub 2012 Jul 18. PMID 22806513
- [Background] Lacy AM, Tasende MM, Delgado S, Fernandez-Hevia M, Jimenez M, De Lacy B, Castells A, Bravo R, Wexner SD, Heald RJ. Transanal Total Mesorectal Excision for Rectal Cancer: Outcomes after 140 Patients. J Am Coll Surg. 2015 Aug;221(2):415-23. doi: 10.1016/j.jamcollsurg.2015.03.046. Epub 2015 Mar 30. PMID 26206640
- [Background] Fernandez-Hevia M, Delgado S, Castells A, Tasende M, Momblan D, Diaz del Gobbo G, DeLacy B, Balust J, Lacy AM. Transanal total mesorectal excision in rectal cancer: short-term outcomes in comparison with laparoscopic surgery. Ann Surg. 2015 Feb;261(2):221-7. doi: 10.1097/SLA.0000000000000865. PMID 25185463
- [Background] Lelong B, de Chaisemartin C, Meillat H, Cournier S, Boher JM, Genre D, Karoui M, Tuech JJ, Delpero JR; French Research Group of Rectal Cancer Surgery (GRECCAR). A multicentre randomised controlled trial to evaluate the efficacy, morbidity and functional outcome of endoscopic transanal proctectomy versus laparoscopic proctectomy for low-lying rectal cancer (ETAP-GRECCAR 11 TRIAL): rationale and design. BMC Cancer. 2017 Apr 11;17(1):253. doi: 10.1186/s12885-017-3200-1. PMID 28399840
- [Background] Hua L, Wang C, Yao K, Zhang J, Chen J, Ma W. Is the incidence of postoperative anastomotic leakage different between laparoscopic and open total mesorectal excision in patients with rectal cancer? A meta-analysis based on randomized controlled trials and controlled clinical trials. J Cancer Res Ther. 2014 Dec;10 Suppl:272-5. doi: 10.4103/0973-1482.151491. PMID 25693934
- [Background] Staudacher C, Vignali A, Saverio DP, Elena O, Andrea T. Laparoscopic vs. open total mesorectal excision in unselected patients with rectal cancer: impact on early outcome. Dis Colon Rectum. 2007 Sep;50(9):1324-31. doi: 10.1007/s10350-007-0289-3. PMID 17665258
- [Background] Veenhof AA, Engel AF, Craanen ME, Meijer S, de Lange-de Klerk ES, van der Peet DL, Meijerink WJ, Cuesta MA. Laparoscopic versus open total mesorectal excision: a comparative study on short-term outcomes. A single-institution experience regarding anterior resections and abdominoperineal resections. Dig Surg. 2007;24(5):367-74. doi: 10.1159/000107778. Epub 2007 Aug 20. PMID 17785982
- [Background] Intention to treat analysis and per protocol analysis: complementary information. Prescrire Int. 2012 Dec;21(133):304-6. PMID 23373104
- [Background] Shah PB. Intention-to-treat and per-protocol analysis. CMAJ. 2011 Apr 5;183(6):696; author reply 696. doi: 10.1503/cmaj.111-2033. No abstract available. PMID 21464181
- [Background] Quirke P, West N. Quality of surgery: has the time come for colon cancer? Lancet Oncol. 2015 Feb;16(2):121-2. doi: 10.1016/S1470-2045(14)71223-9. Epub 2014 Dec 31. No abstract available. PMID 25555422
- See also: Related Info — http://clinicaltrials.gov/ct2/show/NCT02584985
- See also: Related Info — http://www.sealedenvelope.com/power/binary-noninferior/